CLINICAL TRIAL: NCT00842322
Title: The Effect of Increased Fluid Intake on Chronic Renal Failure
Brief Title: Fluid Intake in Kidney Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Martin Haas, MD, Medical University Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OFS1
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Renal Failure; Kidney Transplantation
Keywords: chronic kidney disease; transplantation; kidney function; fluid intake; osmolarity
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fluid intake (Experimental): fluid intake of 4 litres per day
  Interventions: Behavioral: high fluid intake
- normal fluid intake (Experimental): Fluid intake of 2 litres per day
  Interventions: Behavioral: normal fluid intake

INTERVENTIONS:
Behavioral: high fluid intake — fluid intake of 4 litres per day
  Arms: High fluid intake
Behavioral: normal fluid intake — Fluid intake of 2 litres per day
  Arms: normal fluid intake

SUMMARY:
Patients with renal impairment are usually advised to increase their fluid intake. There is currently, however, no evidence supporting this recommendation. In contrast,high fluid intake could be dangerous if urine excretion is reduced. In this study the researchers investigate whether increasing fluid intake from 2 to 4 litres per day has any influence on long-term renal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with native kidney disease or chronic kidney transplant failure
* An effective glomerular filtration rate (eGFR) according the MDRD formula between 20 and 75ml/min/1.73m2
* Ejection fraction >20%
* Absence of liver cirrhosis or ascites
* No evidence of active glomerulonephritis or immunosuppressive therapy if native kidney disease
* Acute transplant rejection
* Urinary protein excretion below 3g/d
* Age between 18 and 70 years.

Exclusion Criteria:

* Therapy resistant edema
* Severe pulmonary disease
* Mean arterial pressure (MAP) > 120 mm Hg
* Pregnancy
* Kidney transplantation within three months prior to randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Haas, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria